CLINICAL TRIAL: NCT06726499
Title: Orthokeratology Lens Decentration with Two Designs of Corneal Refractive Therapy™ Lenses: a One-year Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Gonzalo Carracedo, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16/371-E
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Myopia Progression
Keywords: myopia; orthok
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- spherical design (Experimental)
  Interventions: Device: Spherical CRT
- Toric Design (Experimental)
  Interventions: Device: Toric CRT

INTERVENTIONS:
Device: Spherical CRT — Contact lens for myopia progression
  Arms: spherical design
Device: Toric CRT — Contact lens for myopia progression
  Arms: Toric Design

SUMMARY:
Background/Objectives: To examine the trend of treatment zone (TZ) decentration over 12 months of Orthokeratology (OK) wear using two corneal refractive therapy (CRT) lens designs: standard (STD) and dual axis (DA). Methods: A prospective, randomized, longitudinal study was conducted at the Optometry Clinic of the Complutense University of Madrid. Subjects were fitted with STD or DA designs in one of the eyes, randomly. Refraction, uncorrected visual acuity (VA) and corneal topography were performed at baseline, 1-night, 1-week, 1-, 3-, 6- and 12-month of lens wear. Subjects requiring lens parameter adjustments or replacements after 3 months were excluded. Decentration was measured by subtracting pre-OK from post-OK tangential curvature maps at each visit, with decentration distance and corneal optical TZ measured using MATLAB. Correlations between decentration and visual acuity (VA) were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 to 17 years old
* Myopia up -6.00 D

Exclusion Criteria:

* Ocular diseases

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2018-06-09 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
contact lens centration | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University Complutense of Madrid, Madrid, Madrid, Spain